CLINICAL TRIAL: NCT02148744
Title: A Randomized, Double-Blinded, Placebo-Controlled, Ascending Dose Study of the Safety, Tolerability, and Pharmacokinetics of XmAb®7195
Brief Title: Safety and Tolerability of XmAb®7195 in Adult Healthy Volunteers and Adult Subjects With a History of Allergic Rhinitis and/or Allergic Conjunctivitis and/or Atopic Dermatitis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Xencor, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: XmAb7195-01
Record Dates: First submitted 2014-05-19; First posted 2014-05-28 (Estimated); Last update posted 2017-01-24 (Estimated); Status verified 2017-01

CONDITIONS: Allergic Rhinitis; Allergic Conjunctivitis; Atopic Dermatitis
MeSH Terms: conditions — Rhinitis, Allergic; Conjunctivitis, Allergic; Dermatitis, Atopic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- XmAb7195 or Placebo (Experimental)
  Interventions: Biological: XmAb7195; Biological: Placebo

INTERVENTIONS:
Biological: XmAb7195 — Part 1 and 2: Single IV infusion of XmAb7195 or placebo Part 3: Two-dose sequential IV infusion of XmAb7195 or placebo on Day 1 and Day 8
Biological: Placebo

SUMMARY:
This first-in-human (FIH) study is a randomized, double-blinded, placebo-controlled, ascending dose study to investigate the safety, tolerability, and pharmacokinetics of XmAb7195 in adult healthy volunteers and in adult subjects with elevated IgE levels.

ELIGIBILITY:
Inclusion Criteria:

* Adult males and females 18 to 50 years of age
* Parts 1 and 3: Healthy subjects with no clinically significant abnormality identified on medical or laboratory evaluation and no history of any clinically significant disorder, condition, or disease that would pose a risk to subject safety or interfere with the study evaluation, procedures, or completion;
* Part 2: Otherwise healthy male and female subjects with a history of allergic rhinitis and/or allergic conjunctivitis and/or atopic dermatitis with an elevated serum IgE
* Subjects who are able and willing to give written informed consent;
* Subjects who have the ability to complete all study assessments;
* Subjects who are willing to forego other forms of experimental treatment during the study.

Exclusion Criteria:

* Subjects who have a clinically relevant history or presence of respiratory, gastrointestinal, renal, hepatic, hematological, lymphatic, neurological, cardiovascular, psychiatric, musculoskeletal, genitourinary, immunological, dermatological, connective tissue diseases, or disorders (other than allergic rhinitis and/or conjunctivitis and/or atopic dermatitis in Part 2) that would pose a significant risk to subject safety or significantly interfere with the study evaluation, procedures, or completion
* Subjects who are positive for hepatitis B surface antigen (HBsAg), hepatitis C virus (HCV) antibody and/or human immunodeficiency virus (HIV) Type I or Type II tests at Screening;
* Subjects who do not agree to use medically acceptable methods of contraception (as defined in the protocol);
* Subject is pregnant or breast feeding, or planning to become pregnant within 3 months of administration of XmAb7195;
* Subjects who have used any investigational drug in any clinical trial within 8 weeks prior to admission (Day -1), or have used an experimental monoclonal antibody;
* Subjects with prior exposure to a monoclonal antibody;
* Subjects with a history of anaphylaxis;
* Subjects who have received live vaccines ≤ 3 months from Screening;

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2014-05; Primary Completion 2015-09-21 (Actual); Study Completion 2015-09-21 (Actual)

PRIMARY OUTCOMES:
Number of adverse events including type and severity | Date of randomization up to Day 43
  Number, type and severity of adverse events, vital signs, electrocardiogram (ECGs), laboratory tests, and physical examinations will be reported during the study from randomization up to Day 43
Number of adverse events including type and severity of a priming IV dose followed by an escalating second IV dose | Date of randomization up to Day 36
  Number, type and severity of adverse events, vital signs, electrocardiogram (ECGs), laboratory tests, and physical examinations will be reported during the study from randomization up to Day 36

SECONDARY OUTCOMES:
Blood concentration of XmAb7195 and blood levels of human anti-human antibodies after single-dose IV administration of XmAb7195 | Time of dosing up to Day 43
  Pharmocokinetic (PK) analysis for levels of XmAb7195 will be determined in subjects blood from time of initial dosing up to Day 43
Blood concentration of XmAb7195 and blood levels of human anti-human antibodies after a priming IV dose followed by an escalating second IV dose of XmAb7195 | Time of dosing up to Day 36
  Presence of human anti-human antibodies will be assessed from time of dosing up to Day 36

CONTACTS AND LOCATIONS:
Overall Officials: Ronald Goldwater, MD, Principal Investigator — Parexel Baltimore Early Phase Clinical Unit
Locations (1):
- Parexel Baltimore Early Phase Clinical Unit, Baltimore, Maryland, United States